CLINICAL TRIAL: NCT01158170
Title: A Randomized, Phase III Trial of Prophylactic Cranial Irradiation (PCI) in Patients With Advanced Non-small Cell Lung Cancer (NSCLC) Who Are Effective on Erlotinib or Gefitinib(RT1001)
Brief Title: Prophylactic Cranial Irradiation in Erlotinib/Gefitinib-responders With Non-small Cell Lung Cancer (NSCLC) (RT1001)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Shenglin Ma, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZhejiangCH06
Record Dates: First submitted 2010-06-23; First posted 2010-07-08 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2010-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: nonsmall cell lung cancer; brain metastasis; prophylactic cranial irradiation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Erlotinib Hydrochloride; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prophylactic cranial irradiation (Experimental): Patients receive Erlotinib or gefitinib until disease progression or intolerable toxicity, and prophylactic cranial irradiation 25GY over 10 fractions.
  Interventions: Radiation: Prophylactic cranial irradiation; Drug: Erlotinib /Gefitinib
- Conctrol (Active Comparator): Patients received Erlotinib or gefitinib until disease progression,or intolerable toxicity
  Interventions: Drug: Erlotinib /Gefitinib

INTERVENTIONS:
Radiation: Prophylactic cranial irradiation — 25GY/10fraction
  Other Names: PCI
  Arms: prophylactic cranial irradiation
Drug: Erlotinib /Gefitinib — Erlotinib 150mg/d or Gefitinib 250mg/d until disease progression or intolerable toxicity
  Other Names: EGFR-TKI

SUMMARY:
RATIONALE: Radiation therapy to the brain may be effective in preventing brain metastases in patients with advanced non-small cell lung cancer. It is not yet known whether radiation therapy is more effective than observation in patients with advanced non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying radiation therapy to the brain to see how well it works compared with observation in preventing brain metastases in patients with advanced non-small cell lung cancer

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

Determine the effectiveness of prophylactic cranial radiotherapy in patients with advanced non-small cell lung cancer that is responsive to gefitinib or erlotinib hydrochloride.

Secondary

Determine the progression-free survival in patients treated with this regimen. Determine the overall survival in patients treated with this regimen. Determine the safety and tolerability of this regimen in these patients. Determine the psycho-neurological effects of this regimen in these patients. Determine the quality of life of patients treated with this regimen. OUTLINE: This is a multicenter study. Patients with good response( CR/PR) to EGFR-TKI(Erlotinib or Gefitinib) are randomized to receive EGFR-TKI plus PCI or EGFR-TKI alone,stratified according to prior chemotherapy regimens (first line vs second line), and disease response status.

Group 1: Patients undergo prophylactic brain radiotherapy. Group 2: Patients undergo observation. Patients complete quality of life questionnaires periodically.

After completion of study therapy, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were required to have histologically or cytologically documented
2. NSCLC and no brain metastasis documented by magnetic resonance imaging (MRI)within 21 days after confirmed response (RR+SD) to chemotherapy
3. No previous history of radiotherapy and surgery of brain
4. good response( CR/PR) to Erlotinib or Gefitinib.
5. Agree to radiotherapy
6. age > 18 and <75 years,ECOG performance status 1 or less
7. Good renal and hepatic and haematological (absolute neutrophils count 15 x1O9/L and platelet count 90 x 109/L,HB>=80g /DL) functions
8. Have provided informed consent

Exclusion Criteria:

1. Seizure cannot be controled by the drugs
2. Combined with other disease of the brain such as tumour or infarction
3. Hypersensitivity to MR enhancer -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-05 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the cumulative incidence of symptomatic brain metastases (BM) | 2.5years

SECONDARY OUTCOMES:
overall survival | baseline to date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Shenglin Ma, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China